CLINICAL TRIAL: NCT01747746
Title: Anticoagulation With Rivaroxaban in Post Cardioversion Patients
Brief Title: Anticoagulation With Rivaroxaban in Cardioversion -The ARC Study
Acronym: ARC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cook County Health (Other Government)
Collaborators: Cook County Hospital (Other)
Responsible Party: Principal Investigator, Pete Antonopoulos, Clinical Pharmacist- Principal Investigator, Cook County Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-139
Record Dates: First submitted 2012-11-30; First posted 2012-12-12 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Atrial Fibrillation; Stroke; Thrombo-embolism; Bleeding
Keywords: Rivaroxaban; Warfarin; Anticoagulation; Stroke; Thrombo-embolism; Bleeding; Atrial Fibrillation; Cardioversion
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Hemorrhage | interventions — Rivaroxaban; Warfarin; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Active Comparator): Anticoagulation with Rivaroxaban 20 mg daily with dinner for 30 days
  Interventions: Drug: Rivaroxaban
- Warfarin and Enoxaparin (Other): Warfarin: 1-10 mg per Nomogram Enoxaparin weight based 1 mg/kg Q12 or 1.5 mg/kg/day Historic control
  Interventions: Drug: Warfarin and Enoxaparin

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban versus Historical controlled Anticoagulation with Warfarin and Enoxaparin
  Other Names: Xarelto
  Arms: Rivaroxaban
Drug: Warfarin and Enoxaparin — Historical Control
  Other Names: Coumadin
  Arms: Warfarin and Enoxaparin

SUMMARY:
The purpose of this study is to determine that a new drug called "Rivaroxaban®" is effective in preventing patients from forming clots after their heart rhythm has been reset by the cardiologist with an electrical device.

DETAILED DESCRIPTION:
Patient who are electrically cardioverted require 1 month of anticoagulation (blood thinner). Rivaroxaban a Xa-inhibitor has been shown to be non-inferior to Warfarin (Vit K antagonist) the current standard of care in many treatment areas. Rivaroxaban will be compared to Warfarin historical control group studying the safety and efficacy in electrically cardioverted patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-valvular atrial fibrillation requiring electrical cardioversion o Atrial fibrillation of unknown duration

Exclusion Criteria:

* Patients requiring extended anticoagulation after cardioversion due to concomitant risk factors as defined by CHADS2 score ≥ 1
* Significant renal dysfunction (CrCl <15mL/min)
* Significant hepatic dysfunction (Childs-Pugh Class B or C)
* History of coagulopathy
* Active bleeding
* Hypersensitivity to Rivaroxaban
* Concomitant use of anticoagulants
* Concomitant use of potent CYP3A4/P-gp inhibitors or inducers
* Interventions requiring interruption of therapy
* Pregnancy
* Age <18 y/o
* History of GI Bleed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Thrombosis | 30 days
  Number of cerebrovascular accidents, thrombus and embolism

SECONDARY OUTCOMES:
Mortality | 30 days
  Monitor the 30 day mortality rate
Hospitalizations | 30 days
  Hospitalizations for thrombus or adverse events
Bleeding | 30 days
  The incidence of major and minor bleeding (as defined under 'safety measures')

CONTACTS AND LOCATIONS:
Overall Officials: Pete Antonopoulos, PharmD, Principal Investigator — Cook County Hospital; Asinul Ansari, MD, Principal Investigator — Cook County Hospital
Locations (1):
- Cook County Hospital, Chicago, Illinois, United States